CLINICAL TRIAL: NCT07102797
Title: ActiveGirls: Physical Activity, Hormone Health, and Diabetes Risk in Early Adolescence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rachel Clare Whooten, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2025P001307; 5K23DK131322 (NIH)
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: PCOS (Polycystic Ovary Syndrome); Puberty; Insulin Resistance; Physical Activity
Keywords: PCOS; Prevention; Physical Activity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the intensive intervention group with text messaging and health coaching versus a delayed lower intensity comparison group with a lower intensity text-only intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full Intensity Intervention (Experimental): Participants in this arm will receive the 'full' intensive ActiveGirls intervention, which will include educational messaging (3-4/week, via email or text message) as well as a series of 6 health coaching visits for physical activity goal setting. Participants in this arm will receive the intervention in months 1-6 of their study participation.
  Interventions: Behavioral: ActiveGirls Physical Activity Program (Full)
- Delayed lower intensity comparison group (Active Comparator): Participants in this arm will receive a lower intensity educational messaging only intervention in months 7-12 of their study participation. This group will not receive health coaching.
  Interventions: Behavioral: ActiveGirls Physical Activity Program (Delayed Lower Intensity)

INTERVENTIONS:
Behavioral: ActiveGirls Physical Activity Program (Full) — Participants in the ActiveGirls Full Intensity intervention group will receive a series of 6 health coaching visits delivered via telemedicine. These visits will address physical activity goal setting within the family. Participants will also receive the ActiveGirls education messaging which will include 3-4 text messages per week (Months 1-6 of their study participation).
  Arms: Full Intensity Intervention
Behavioral: ActiveGirls Physical Activity Program (Delayed Lower Intensity) — Participants in this group will only receive the ActiveGirls education messaging which will include 3-4 text messages per week (Months 7-12 of their study participation)
  Arms: Delayed lower intensity comparison group

SUMMARY:
This study explores how a physical activity program can affect hormone health and diabetes risk in girls ages 8-12 who may be at higher risk. The study aims to address:

* Does the 'ActiveGirls' program meet the needs of girls and families in engaging them to increase physical activity?
* What is the trend of markers of diabetes risk and puberty hormones over a 1-year period and how are these levels related to physical activity levels?

Participants in this study will either:

* Participate in a 'full' intensity intervention that includes educational messages (text/email) as well as health coaching visits to support physical activity over a 6 month period
* Participate in a delayed 'lower intensity' intervention that includes only educational messages (text/email)
* Participants in both groups will complete at-home activity monitoring, two study visits for check-ups and tests, and surveys

DETAILED DESCRIPTION:
This study is a pilot randomized trial to assess the preliminary feasibility and efficacy of a physical activity intervention enrolling peripubertal females.

Participants will be assigned to the intensive intervention group with text messaging and health coaching versus delayed lower intensity comparison group with a lower intensity text-only intervention. Participants in both arms will complete objective measures of body composition, insulin dynamics, reproductive hormones, physical activity and fitness over a one-year period. Participants as well as a caregiver proxy will complete survey measures addressing lifestyle behaviors and social-emotional wellness. Given evidence suggesting increased effectiveness of whole-family lifestyle interventions, a parent/caregiver will assist with child participation in the ActiveGirls program, including facilitating health coaching visits and at-home physical activity sessions. assist in intervention delivery and outcomes assessment.

After the baseline visit, there are 2 more study assessment points at 6-months and 12-months. The baseline and 12-month assessments require in-person visits to the MGH Translational and Clinical Research Centers (TCRC); the 6-month assessment is performed remotely. All study visits will occur at MGH.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver: Caregiver of child (ie mother, father, or other legal guardian), English-speaking, Access to a device where they are able to receive study e-mails or texts
* Child: English-speaking, Female, ages 8-12 years old at time of enrollment, Pre-menarchal at time of baseline visit, at risk for Polycystic Ovary Syndrome (PCOS)/insulin resistance, as defined by (1) History of maternal PCOS/maternal GDM, (2) BMI >/= 85th percentile, (3) History of premature adrenarche, or (4) Small (<10th %ile) for gestational age

Exclusion Criteria (Child):

* Medications at time of enrollment: Metformin, GLP-1R Agonist, Insulin, GnRH agonist
* Endocrine conditions that would impact either insulin sensitivity, androgen concentrations, or growth
* Insulin dynamics: Type 1 diabetes, Type 2 diabetes, Congenital Hyperinsulinism
* Androgen Conditions: Adrenal tumor, Congenital Adrenal Hyperplasia
* Hyperthyroidism or uncontrolled hypothyroidism (TSH >7.0 mIU/mL)
* Growth Hormone Deficiency
* Medical conditions that would impact PA participation: Type 1 diabetes; Cardiovascular, neurologic, and/or musculoskeletal conditions limiting ability to participate in physical activity.
* Other medical comorbidities that would limit generalizability of findings, including: Severe congenital heart disease, Congenital anomalies, Cystic fibrosis, Cerebral palsy, Condition requiring use of nasogastric, gastric tube, or other alternative method of feeding, Undiagnosed conditions with significant impact on child's growth and development; Significant cardiac, hepatic, oncologic, inflammatory, or psychiatric disease.

Min Age: 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Retention | 12 months
  Proportion of participants completing each study assessment point/coaching visit divided by total participants enrolled/eligible
Acceptability | 12 months
  Intervention rating as acceptable by parent-child dyads using validated measure (Acceptability of Intervention Measure (AIM)); The AIM score is reported on a scale of 0-4. 0 is the minimum and 4 is the maximum. Higher scores mean greater intervention acceptability

SECONDARY OUTCOMES:
Objectively Measured Physical Activity | 6 months, 12 months
  Change in MVPA (minutes/day) from baseline to 6-month and 12-month follow-up
Insulin Sensitivity | Change in HOMA-IR from baseline to 12-month follow-up
  As measured by HOMA-IR (unitless; calculated based on product of fasting insulin and fasting glucose using standardized formula)
Free Androgen Index | Baseline to 12 month follow-up
  Calculated using Total Testosterone and SHBG

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided